CLINICAL TRIAL: NCT05639244
Title: Effect of Short Term Time Restricted Eating on Innate Immunity in Patients With Coronary Artery Disease
Brief Title: Time Restricted Eating and Innate Immunity
Acronym: SIGNATURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NL80950.091.22
Record Dates: First submitted 2022-10-16; First posted 2022-12-06 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-11

CONDITIONS: Time Restricted Feeding; Myocardial Infarction; Atherosclerotic Cardiovascular Disease
Keywords: time restricted eating
MeSH Terms: conditions — Intermittent Fasting; Myocardial Infarction; Atherosclerosis | interventions — Diet

STUDY DESIGN:
Intervention Model Description: The investigators will include 20 adult patients. Participants will be randomised to a 2 week time restricted eating (TRE) period or a 2 week period in which they consume their regular diet within an unrestricted time period. Participants will be crossed over to the other treatment arm after a 6 weeks wash-out period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First TRE, then regular diet (Other): This group will start with 2 weeks TRE and will switch to the 2 week period of consuming their regular diet after a wash-out period.
  Interventions: Behavioral: Time restricted eating (TRE); Behavioral: Regular diet
- First regular diet, then TRE (Other): This group will start with the 2 week period of consuming their regular diet and will switch to 2 weeks TRE after a wash-out period.
  Interventions: Behavioral: Time restricted eating (TRE); Behavioral: Regular diet

INTERVENTIONS:
Behavioral: Time restricted eating (TRE) — Participants have to consume their regular food intake during a 6 hour period per day for 2 weeks.
Behavioral: Regular diet — Participants have to consume their regular diet within an unrestricted time period for 2 weeks

SUMMARY:
The goal of this cross over study is to investigate the effect of short term time restricted eating (TRE) on the innate immune system in patients with a history of myocardial infarction.

DETAILED DESCRIPTION:
In the recent years, research has shown the prominent role of low grade systemic inflammation in cardiovascular disease (CVD) and the crucial role myeloid cells, mainly monocytes and macrophages, play in atherogenesis. Time restricted eating (TRE), i.e. eating the normal amount of calories within a limited time period per day, has a beneficial effect on multiple factors involved in the development of CVD, such as blood pressure, heart rate, lipid and blood glucose levels, and insulin sensitivity. TRE also reduces markers of systemic inflammation and reduces the number of circulating monocytes.

It is now hypothesized that TRE reduces the pro-inflammatory monocyte phenotype of patients with a history of myocardial infarction. Therefore, the investigators will perform a exploratory prospective randomised open label blinded endpoint cross-over study to investigate the effect of short term TRE on the innate immune system in patients with a history of myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age >18 years)
* Diagnosed with a myocardial infarction (between 1 and 5 years ago)
* Body mass index between 20 and 35 kg/m2
* Able to understand, be motivated and follow the study related procedures
* Able to understand and give written informed consent

Exclusion Criteria:

* Myocardial infarction (defined as an increase in cardiac enzymes in combination with symptoms of ischemia or newly developed ischemic ECG changes), coronary artery bypass graft surgery or other major (cardiovascular) surgery, stroke or transient ischemic attack (TIA) in the past 1 year prior to screening.
* Use of immunomodulatory drugs
* Use of drugs that need to be taken with food.
* Diabetes Mellitus type I and type II
* Medical history of any disease associated with immune deficiency (either congenital or acquired, including chemotherapy, active malignancy, organ transplant) or auto immune disease
* Clinically significant infections within 1 months prior to start of or during intervention period or control period (defined as fever >38.5).
* Vaccination <1 month before start of or during intervention or control period.
* Eating disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
The change in the inflammatory phenotype of circulating immune cells, assessed by measuring the cytokine production capacity (e.g. IL-1b and TNF) of isolated PBMCs after ex vivo stimulation with various TLR ligands, determined by ELISA. | Change from baseline cytokine production capacity at 2 weeks after TRE or regular diet.
  The investigators will measure the change in the inflammatory phenotype of circulating immune cells after TRE.
  Therefore, the investigators will assess the inflammatory phenotype at baseline and after a two week TRE period and a control period with a regular diet (cross-over design).
  This will be assessed by measuring the cytokine production capacity of isolated peripheral blood mononuclear cells (PBMCs) after ex vivo stimulation with various TLR ligands. Relevant cytokines (e.g. IL-1b and TNF, given in pg/ml) are measured in the supernatants of the PMBC stimulation experiments by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Niels P. Riksen, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be published in a data repository or other online data archive (e.g. DANS EASY, Radboud Data Repository, disciplinary repository, data archive). Data that is applicable for sharing (regarding privacy) will be published.
Time Frame: All data from the research project will be shared after the publication of the results.
Access Criteria: All data will be made available without restrictions.